CLINICAL TRIAL: NCT04948983
Title: Patient Decision Aids for Women Facing the Decision of Breast Cancer Screening in the Public Health Sector
Brief Title: The Effect of a Patient Decision Aids for Breast Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SA18i0002
Record Dates: First submitted 2021-06-07; First posted 2021-07-02 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Mammary Cancer; Breast Tumor; Mammary Tumor
Keywords: Breast Cancer; Decision aid; Decision making process; Mammography; Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: The intervention group will access a webpage, answers a set of questionnaires at baseline, and then the DA (developed according to the IPDAS recommendations). The Control group will access a webpage, answers a set of questionnaires at baseline, and then receive standardised information given by the healthcare system. Both groups will complete the questionnaires two weeks later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will access a web page, answer a set of questionnaires at baseline, and then the DA (developed according to the IPDAS recommendations). The intervention group will complete the same questionnaires two weeks later. Six months later we will confirm if the screening was undertaken by checking medical records.
  The online DA for breast cancer screening is a web-based education material to inform women about the benefits and risks associated with the screening. The contents of the DA are: 1) Assessing breast cancer; 2) What is breast cancer screening?; 3) What will happen if I diagnosed with breast cancer?; 4) What is overdiagnosis?; 5) What is false positive?; 6) the statistics of breast cancer screening; 7) Now is my turn, do I want to take it?
  Interventions: Other: Decision aid (DA) for breast cancer screening
- Control group (Placebo Comparator): The Control group will access a webpage, answer a set of questionnaires at baseline, and then receive standardised information given by the healthcare system.
  The control group will complete the same questionnaires two weeks later, afterwards they will access the DA. Six months later we will confirm if the screening was undertaken by checking medical records.
  Interventions: Other: Standarised information for breast cancer screening

INTERVENTIONS:
Other: Decision aid (DA) for breast cancer screening — The online DA for breast cancer screening is a web-based education material to inform women about the benefits and risks associated with the screening. The contents of the DA are: 1) Assessing breast cancer; 2) What is breast cancer screening?; 3) What will happen if I diagnosed with breast cancer?; 4) What is overdiagnosis?; 5) What is false positive?; 6) the statistics of breast cancer screening; 7) Now is my turn, do I want to take it?
  Arms: Intervention group
Other: Standarised information for breast cancer screening — Information provided by the Chilean Ministry of Health in regards to access to breast cancer screening (Age, frequency and costs)
  Arms: Control group

SUMMARY:
Breast cancer is one of the most common cancers in Chile. National efforts focus on early detection, offering universal access to breast cancer screening through mammography to women at risk age. However, 30% of women do not undertake the exam due to a lack of knowledge and anxiety when facing the decision. The aim of this study is to develop and evaluate the effectiveness of a decision aid (DA) for women facing breast cancer screening decision in the country. Methods: following the Medical Research Council guidelines for the development and implementation of a complex intervention in public health, the investigators have: 1) culturally adapted the German DA for mammography; 2) conducted focus groups with experts to further develop the DA; 3) pilot-tested the online DA with 20 women in primary care centres.

A total of 3,269 women aged 50 to 69 years old are invited to join the study. The intervention group accesses a webpage, answers a set of questionnaires at baseline, and then the DA (developed according to the IPDAS recommendations). The Control group accesses a webpage, answers a set of questionnaires at baseline, and then receives standardised information given by the healthcare system. Both groups complete the questionnaires two weeks later. The primary outcome measure is an adapted and validated version of Informed Choice. Additionally, decisional conflict, anxiety, and screening undertake rate are measured. Multiple lineal regression analysis will be conducted.

DETAILED DESCRIPTION:
There is an alarming rise of breast cancer in developing countries, where early detection is rare and the late findings build up an important mortality rate. In Chile, the mortality rate is 15,5 per 100.000 women, where breast cancer is the first death caused by tumors. Governmental efforts had focused on increase an opportune detection and had offered universal and guaranteed access to breast cancer screening to women in at-risk age (50 to 59 years old). Still, about 30% of the women of at-risk age choose to not do the mammogram. Anxiety and lack of awareness are the principal reasons associated with the decision of rejecting or postponing the exam. Women would have trouble in making an informed decision about the breast cancer exam, resulting in possible negatives consequences for their wellbeing. Considering that the health-related decision-making process depends importantly on the personal balance of risk and benefits related to the decision, it is imperative to explore strategies that support women in the decision-making progress for breast cancer screening.

The aim of this study is to develop and evaluate the effectiveness of a decision aid (DA) for women facing breast cancer screening decision in the country. Methods: following the Medical Research Council guidelines for the development and implementation of a complex intervention in public health, the investigators have: 1) culturally adapted the German DA for mammography; 2) conducted focus groups with experts to further develop the DA; 3) pilot-tested the online DA with 20 women in primary care centres; 4) A two-arm randomized control trial will be conducted with a total of 3,269 women aged 50 to 69 years old in ten primary care centres in Chile.

The intervention group will access a webpage, answers a set of questionnaires at baseline, and then the DA (developed according to the IPDAS recommendations). The Control group will access a webpage, answers a set of questionnaires at baseline, and then receives standardised information given by the healthcare system. Both groups will complete the questionnaires two weeks later. The primary outcome measure is an adapted and validated version of Informed Choice. Additionally, decisional conflict, anxiety, and screening undertake rate will be measure. Multiple lineal regression analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Women from 50 to 69 years old
* Attend the primary care centres
* Fluent in Spanish

Exclusion Criteria:

* Women with a personal history of breast cancer
* Have a current mammogram (as recommended by the Chilean Ministry of Health)
* Not having the capacity to consent.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3269 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Informed choice for breast cancer screening | Change from baseline informed choice at two weeks
  An adapted and validated version of the informed choice questionnaire will be used: this is a five-item questionnaire to measure informed choice (Bravo P, Dois A, Fernández-González L, Hernández-Leal MJ, Villarroel L. [Validation of the Informed Choice instrument for Chilean women facing a mammography decision in primary care]. Aten Primaria. 2021 Mar;53(3):101943. doi: 10.1016/j.aprim.2020.08.005. Epub 2021 Feb 13. Spanish. PubMed ID: 33592532).
  Minimum value= 5 Maximum value= 25

SECONDARY OUTCOMES:
Decisional conflict | Change from baseline decisional conflict at two weeks
  Decisional conflict scale with 16 items that measure uncertainty in the decision making process.
  Minimum value= 16 Maximum value= 80
Depression, anxiety and stress | Change from baseline drepression, anxiety and stress at two weeks
  This will be measured with the DASS-21 Scale, a self-reported 21-item that captures depression, anxiety and stress during the last week.
  Minimum value= 21 Maximum value= 84
Satisfaction with the decision | Change from baseline satisfaction with the decision at two weeks
  This is a two-item self-reported satisfaction questionnaire related to breast cancer screening.
  Minimum value= 0 Maximum value= 1
Number of participants who undertake a mammography | At 6 months
  This will be the number of women who decided to undertake the mammography. This outcome will be obtained from the clinical record of each participant six months after baseline questionnaires.
  Minimum value= 0 Maximum value= 1

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Bravo, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Alejandra Martínez, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bravo P, Dois A, Fernandez-Gonzalez L, Hernandez-Leal MJ, Villarroel L. [Validation of the Informed Choice instrument for Chilean women facing a mammography decision in primary care]. Aten Primaria. 2021 Mar;53(3):101943. doi: 10.1016/j.aprim.2020.08.005. Epub 2021 Feb 13. Spanish. PMID 33592532
- [Derived] Riganti P, Ruiz Yanzi MV, Escobar Liquitay CM, Sgarbossa NJ, Alarcon-Ruiz CA, Kopitowski KS, Franco JV. Shared decision-making for supporting women's decisions about breast cancer screening. Cochrane Database Syst Rev. 2024 May 10;5(5):CD013822. doi: 10.1002/14651858.CD013822.pub2. PMID 38726892